CLINICAL TRIAL: NCT05355584
Title: Acute Effects of Cryotherapy Duration on Muscle Strength, Flexibility, Endurance and Balance in Healthy Individuals
Brief Title: Acute Effects of Cryotherapy Duration in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burcu Camcıoğlu Yılmaz (Other)
Responsible Party: Sponsor-Investigator, Burcu Camcıoğlu Yılmaz, PT, PhD, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KPR2
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Cryotherapy Effect
Keywords: Cryotherapy; Muscle strength; Flexibility; Endurance; Balance; Healthy people; Cold pack; Shoulder

STUDY DESIGN:
Intervention Model Description: Individuals aged 18-25 years who volunteer to participate in the study will be included in this study and randomly assigned to 3 groups. After the demographic information of the volunteers is obtained and their dominant upper extremities are determined, the shoulder isometric muscle strength will be measured with a hand dynamometer. The back scratch test will be used to evaluate the shoulder flexibility of the participants, the modified push-up test will be used to evaluate the endurance, and the upper extremity Y balance test will be used to evaluate the shoulder dynamic balance. Then, cryotherapy will be applied on the shoulder for 10 minutes in Group 1, 15 minutes in Group 2 and 20 minutes in Group 3.After the application, the same measurements will be repeated and the values before and after the application will be compared.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10-minute Cryotherapy Application (Active Comparator): A cold application will be made on the shoulder for 10 minutes. Before and after the application, individuals will be evaluated in terms of muscle strength, flexibility, endurance and balance. The values before and after the application will be compared.
  Interventions: Other: Cryotherapy application
- 15-minute Cryotherapy Application (Active Comparator): A cold application will be made on the shoulder for 15 minutes. Before and after the application, individuals will be evaluated in terms of muscle strength, flexibility, endurance and balance. The values before and after the application will be compared.
  Interventions: Other: Cryotherapy application
- 20-minute Cryotherapy Application (Active Comparator): A cold application will be made on the shoulder for 20 minutes. Before and after the application, individuals will be evaluated in terms of muscle strength, flexibility, endurance and balance. The values before and after the application will be compared.
  Interventions: Other: Cryotherapy application

INTERVENTIONS:
Other: Cryotherapy application — The temperature sense test was applied on the dominant side shoulder of the participants against the risk of sensory loss or decreased sensation. In order to test cold intolerance, a cold pack was placed on the forearm of the individuals. After waiting 2-3 minutes, the region was evaluated. Individuals meeting the inclusion criteria were assigned to the groups according to the randomization list created by the computer. Then, the participants' shoulder isometric muscle strength, shoulder flexibility, shoulder endurance and shoulder balance was evaluated. Except for shoulder endurance, all measurements were repeated three times, with a 30-second rest period between each repetition. A 2-3-minute rest period was given after each test. Then, the cold pack was wrapped in a thin and wet cloth on the shoulders of the participants. The treated area was checked every 5 minutes and the participants were asked to say when they felt any unusual symptoms.

SUMMARY:
The study will investigate the acute effects of cryotherapy duration on shoulder muscle strength, flexibility, endurance and dynamic balance in healthy individuals.

DETAILED DESCRIPTION:
Cryotherapy is a practice that induces therapeutic effects by reducing tissue temperature to produce an analgesic effect. Cryotherapy application methods vary from simple ice packs and cold water immersion to whole body cryotherapy methods. The purpose of cryotherapy treatment is to reduce tissue damage, muscle spasm, edema and pain and to provide a faster rehabilitation process after injury. It is also used as a recovery technique after high-intensity training in different sports branches. Despite the proven benefits of cryotherapy according to the literature, discussions continue about its effect on some parameters and there is no consensus on the duration of cryotherapy application. In addition, although there are studies on the effects of cryotherapy on the lower extremities, studies for the upper extremity are limited and the results of these studies are inconsistent. In the literature, no study was found that evaluated the effect of cryotherapy application time on shoulder muscle strength, endurance, flexibility and balance. Therefore, in this study, the acute effects of cryotherapy duration on shoulder muscle strength, flexibility, endurance and dynamic balance in healthy individuals will be investigated and the optimum duration of cryotherapy on these parameters will be determined. In addition, the results of the research will contribute to the planned rehabilitation and exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-25 who volunteer to participate in the study
* No upper extremity orthopedic problems
* No history of shoulder injury or surgery in the past two years
* Absence of Raynaud's disease or cold intolerance

Exclusion Criteria:

* Having a history of shoulder injury or surgery
* Cervical or thoracic spine disorders
* People with any neurological disorder or known balance/proprioceptive deficits
* Decreased sensation or decreased blood flow
* Have Raynaud's disease or any cold intolerance

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Muscle Strength | Just before and within 5 minutes after cryotherapy cryotherapy
  Isometric strength of shoulder flexors, extensors, abductors, adductors, internal and external rotators will be measured with a hand dynamometer and recorded in kg. Each muscle group will be tested in three repetitions according to the procedures described by Kendall et al. The average of the three scores will be used for analysis.
Change in Shoulder Flexibility | Just before and within 10 minutes after cryotherapy
  It will be evaluated with the Back Scratch Test. In this test, while in a standing position, the person's fingers are extended (stretched) and the arm is rotated outward with the palm facing the back, towards the ground over the shoulder and while doing this, the other arm is internally rotated, with the palm facing forward and the fingers extended. The distance between the middle fingers of both hands will be measured. If the middle fingers do not touch, the distance between them is recorded as (-) in cm, if the middle fingers touch end to end, the value is (0), if the middle finger crosses the other, the distance between the middle finger is recorded as (+) in cm. Keith et al. reported that the test had a high reliability coefficient (left hand, rxy=0.77 and right hand rxy=0.75).
Change in Shoulder Functional Balance | Just before and within 10 minutes after cryotherapy
  The Y Balance Test kit will be used in the medial, superolateral and inferolateral directions with an angle of 135-135-90 degrees between them. While the dominant hand on the test kit is in the push-up position with the hand at the junction of the angles, the farthest point that the participants can reach with the fingertip of the other hand. and the distance he can reach will be measured in cm.
Change in Shoulder Muscle Endurance | Just before and within 15 minutes after cryotherapy
  Modified Push-up Test will be used. In the test, individuals are positioned face down on the mat with their knees and elbows flexed. The participant will be asked to push his torso backwards by extending his elbows without disturbing the flexion of the knees. The number of correct moves in 30 seconds will be recorded.

SECONDARY OUTCOMES:
Temperature Sensation | Before cryotherapy
  The test will be performed on the shoulder with eyes closed, by putting hot water (40-45 degrees) in one of two glass tubes of equal diameter and cold water (5-10 degrees) in the other. Then, these tubes will be touched to the person and the person will be asked to tell which is hot and which is cold.
Cold Intolerance | Before cryotherapy
  There are four types of symptoms in cold intolerance: pain/discomfort, stiffness, dysesthesia (numbness or tingling), and discoloration. In order to test cold intolerance, cold application will be made on the forearm of the individuals and waited for 2-3 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Camcıoğlu Yılmaz, PT,PhD, Study Director — Muğla Sıtkı Koçman University; Ferhan Beril Yıldız, MSc. Student, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman University Training and Research Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Algafly AA, George KP. The effect of cryotherapy on nerve conduction velocity, pain threshold and pain tolerance. Br J Sports Med. 2007 Jun;41(6):365-9; discussion 369. doi: 10.1136/bjsm.2006.031237. Epub 2007 Jan 15. PMID 17224445
- [Background] Swenson C, Sward L, Karlsson J. Cryotherapy in sports medicine. Scand J Med Sci Sports. 1996 Aug;6(4):193-200. doi: 10.1111/j.1600-0838.1996.tb00090.x. PMID 8896090
- [Background] Bleakley C, McDonough S, MacAuley D. The use of ice in the treatment of acute soft-tissue injury: a systematic review of randomized controlled trials. Am J Sports Med. 2004 Jan-Feb;32(1):251-61. doi: 10.1177/0363546503260757. PMID 14754753
- [Background] Costello JT, Baker PR, Minett GM, Bieuzen F, Stewart IB, Bleakley C. Whole-body cryotherapy (extreme cold air exposure) for preventing and treating muscle soreness after exercise in adults. Cochrane Database Syst Rev. 2015 Sep 18;2015(9):CD010789. doi: 10.1002/14651858.CD010789.pub2. PMID 26383887
- [Background] Bleakley CM, Costello JT, Glasgow PD. Should athletes return to sport after applying ice? A systematic review of the effect of local cooling on functional performance. Sports Med. 2012 Jan 1;42(1):69-87. doi: 10.2165/11595970-000000000-00000. PMID 22121908
- [Background] Rowsell GJ, Coutts AJ, Reaburn P, Hill-Haas S. Effect of post-match cold-water immersion on subsequent match running performance in junior soccer players during tournament play. J Sports Sci. 2011 Jan;29(1):1-6. doi: 10.1080/02640414.2010.512640. PMID 21077001
- [Background] Wilcock IM, Cronin JB, Hing WA. Water immersion: does it enhance recovery from exercise? Int J Sports Physiol Perform. 2006 Sep;1(3):195-206. doi: 10.1123/ijspp.1.3.195. PMID 19116434
- [Result] Keith NR, Clark DO, Stump TE, Miller DK, Callahan CM. Validity and reliability of the Self-Reported Physical Fitness (SRFit) survey. J Phys Act Health. 2014 May;11(4):853-9. doi: 10.1123/jpah.2012-0264. Epub 2013 May 10. PMID 23676451
- [Result] Gorman PP, Butler RJ, Plisky PJ, Kiesel KB. Upper Quarter Y Balance Test: reliability and performance comparison between genders in active adults. J Strength Cond Res. 2012 Nov;26(11):3043-8. doi: 10.1519/JSC.0b013e3182472fdb. PMID 22228174
- [Result] Borms D, Maenhout A, Cools AM. Upper Quadrant Field Tests and Isokinetic Upper Limb Strength in Overhead Athletes. J Athl Train. 2016 Oct;51(10):789-796. doi: 10.4085/1062-6050-51.12.06. Epub 2016 Nov 11. PMID 27834503
- [Result] Campbell DA, Kay SP. What is cold intolerance? J Hand Surg Br. 1998 Feb;23(1):3-5. doi: 10.1016/s0266-7681(98)80207-6. PMID 9571469